CLINICAL TRIAL: NCT06201364
Title: External Oblique Intercostal Block Versus Paravertebral Block for Postoperative Analgesia in Laparoscopic Cholecystectomy Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Adel Abdelkareem, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: External oblique intercostal
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI group (Experimental): chest wall will be systematically scanned. Initially the probe will be placed in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle will be identified at the level ribs 6 and 7 in line with the xiphoid process to confirm correct identification of the external oblique muscle, the probe will be moved in the caudad direction following the external oblique muscle. At the subcostal level, the ultrasound probe will be rotated 90° to see the convergence with the internal oblique and transversus abdominus muscles. The probe will be then moved back to the initial identification point for the external oblique muscle. The EOI plane will be identified deep to the external oblique muscle and superficial to the sixth and seventh ribs and their associated intercostal muscles. Local anesthetic agent will be 20 ml volume (10 ml bupivacaine 0.5% ,10ml saline) will be then injected, this procedure will be done bilaterally.
  Interventions: Procedure: The external oblique intercostal block
- PVB group (Active Comparator): we will be scanning the anatomy of the lateral paravertebral space using a high-frequency linear ultrasound transducer, after identification of the transverse process, internal intercostal membrane (IIM), and pleura at the T3 and T6 levels, an out-of-plane needle guidance technique would be used to perform the PVB with 20 ml volume (10 ml bupivacaine 0.5% ,10ml saline) will be then injected, this procedure will be done bilaterally.
  Interventions: Procedure: Paravertebral block

INTERVENTIONS:
Procedure: The external oblique intercostal block — chest wall will be systematically scanned. Initially the probe will be placed in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle will be identified at the level ribs 6 and 7 in line with the xiphoid process to confirm correct identification of the external oblique muscle, the probe will be moved in the caudad direction following the external oblique muscle. At the subcostal level, the ultrasound probe will be rotated 90° to see the convergence with the internal oblique and transversus abdominus muscles. The probe will be then moved back to the initial identification point for the external oblique muscle. The EOI plane will be identified deep to the external oblique muscle and superficial to the sixth and seventh ribs and their associated intercostal muscles. Local anesthetic agent will be 20 ml volume (10 ml bupivacaine, 10 ml saline) will be injected under ultrasound guidance and this will be done bilaterally.
  Arms: EOI group
Procedure: Paravertebral block — involve injection of local anaesthetic in a space immediately lateral to where the spinal nerves emerge from the intervertebral foramina. This technique is being used increasingly for not only intra-operative and post-operative analgesia but also as a sole anaesthetic technique for carrying out various procedures.
  Arms: PVB group

SUMMARY:
To compare external oblique intercostal block versus paravertebral block for post operative analgesia in patients undergoing laparoscopic cholecystectomy to decease post operative opioid consumption and use the least dose of local anesthesia.

DETAILED DESCRIPTION:
Paravertebral Block (PVB) involve injection of local anesthetic in a space immediately lateral to where the spinal nerves emerge from the intervertebral foramina. This technique is being used increasingly for not only intra-operative and post-operative analgesia but also as a sole anesthetic technique for carrying out various procedures. This popularity is mainly due to the ease of the technique and fewer complications.

The external oblique intercostal block is a novel motor- and opioid-sparing technique which blocks both the anterior and lateral cutaneous branches of the thoracoabdominal nerves which innervate the upper abdominal quadrant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20-60 years old
* Patients with ASA clinical status I\II
* Patients schedule for laparoscopic cholecystectomy

Exclusion Criteria:

* Patients refusal
* Coagulopathy
* Infection at site of injection
* Allergy of local anesthesia
* Sever cardiac disease
* Patients with chest wall deformities

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
total morphine consumption | first 24 hours postoperatively

SECONDARY OUTCOMES:
Time of first rescue analgesia | hours
  rescue analgesia will be given in the form of morphine 4 mg when VAS score ≥4
Visual analogue scale (VAS) | at 0.5 ,1,2,4,8,12,24 hours postoperatively
  It is a validated subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

IPD SHARING:
Plan to Share IPD: Undecided